CLINICAL TRIAL: NCT05347069
Title: Efficacy and Safety of Aspirin in Patients With Chronic Coronary Syndromes Without Revascularization
Acronym: ASA-IN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Takeshi Morimoto (Other)
Responsible Party: Sponsor-Investigator, Takeshi Morimoto, Study Statistician, Kyoto University, Graduate School of Medicine
Organization: Kyoto University, Graduate School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Y0126
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Stable Angina Pectoris; Coronary Artery Disease; Ischemic Heart Disease
Keywords: Chronic Coronary Syndrome; Aspirin
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease; Myocardial Ischemia | interventions — Aspirin; N-acetyl-S-(alpha-methyl-4-(2-methylpropyl)benzeneacetyl)cysteine 4-(nitrooxy)butyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin (Active Comparator): Aspirin 100 mg/day
  Interventions: Drug: Aspirin
- No Aspirin (Active Comparator): No Aspirin
  Interventions: Drug: No aspirin

INTERVENTIONS:
Drug: Aspirin — Aspirin 100 mg/day
  Arms: Aspirin
Drug: No aspirin — No aspirin administered
  Arms: No Aspirin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety aspirin in patients with chronic coronary syndromes without revascularization.

DETAILED DESCRIPTION:
Aspirin for secondary prevention in the acute phase of acute coronary syndromes has been established. Although it is still disputable about the duration, there is also a consensus for antiplatelet therapy in patients after percutaneous coronary revascularization. On the other hand, several large randomized clinical trials (RCTs) have shown that aspirin treatment for primary prevention of cardiovascular events increases bleeding events and does not provide net clinical benefit.Patient with chronic coronary syndromes (CCS) but not eligible for revascularization do not belong to any of these categories and there is no evidence on the efficacy of aspirin in this population. Therefore, we designed a multicenter, randomized, open-label study to evaluate the efficacy and safety of aspirin in patients with CCS who are not eligible for revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic coronary syndromes with ≧50% diameter stenosis in one or more major coronary vessels/major branches on coronary CT or coronary angiography but not eligible for coronary revascularization
* Patients for whom consent can be obtained

Exclusion Criteria:

* Patients with history of acute coronary syndromes (ACS)
* Patients with history of percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)
* Patients with left main trunk stenosis (≥50%)
* Patients for whom aspirin administration is mandatory
* Patients undergoing antithrombotic therapy other than aspirin
* Patients with atrial fibrillation
* Patients with history of stroke within six months
* Patients scheduled for major surgical procedures that will require aspirin discontinuation
* Patients with contraindication of aspirin
* Patients expected to have a prognosis of 1 year or less due to comorbidities
* Women of child-bearing potential or women who have a positive pregnancy test at enrolment or randomization
* Patients who are judged by attending physicians to be inappropriate to participate in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2890 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Composite cardiovascular events | 5 years
  Composite of all-cause death, myocardial infarction, ischemic stroke, coronary revascularization, peripheral revascularization, or critical limb ischemia

SECONDARY OUTCOMES:
All-cause death | 5 years
  As classified by Academic Research Consortium (ARC) (Circulation. 2007;115:2344-2351).
  1. Cardiac Death: Any death due to proximate cardiac cause, unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment. All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in subjects with coexisting potentially fatal non-cardiac disease should be classified as cardiac.
  2. Vascular Death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  3. Non-cardiovascular Death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  4. Cancer related death: death from cancer cause
Myocardial infarction | 5 years
  As classified by Academic Research Consortium (ARC): However, the sensitivity is too high for the evaluation with Troponin of the peri-procedural MI, thus CKMB will be used.
Ischemic stroke | 5 years
  Ischemic stroke is defined as acute onset of a neurological deficit that persists for at least 24 hours and is the result of a disturbance of the cerebral circulation due to ischemia. Deficits that last ≤ 24 hours are due to transient ischemic neurological attack and are not classified in this category.
Coronary revascularization | 5 years
  The revascularization that meets the following criteria is considered as clinically indicated revascularization. Presence/absence of clinical findings is judged by the operator of the procedure before the revascularization.
Peripheral revascularization | 5 years
  The revascularization that meets the following criteria is considered as clinically indicated revascularization. Presence/absence of clinical findings is judged by the operator of the procedure before the revascularization.
Critical limb ischemia | 5 years
  Critical limb ischemia is defined by chronic ischemic pain at rest and/or presence of ischemic skin lesions (gangrene or ulcerations).
Cardiovascular death | 5 years
  1. Cardiac Death: Any death due to proximate cardiac cause (e.g. myocardial infarction [MI], low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment. All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in subjects with coexisting potentially fatal non-cardiac disease (e.g. cancer, infection) should be classified as cardiac.
  2. Vascular Death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
Major bleeding | 5 years
  Bleeding/Hemorrhagic Complications will be evaluated using the Bleeding Academic Research Consortium (BARC) definition. Major bleeding is defined as BARC 3 or 5.
Hospital admission for heart failure | 5 years
  An unplanned hospitalization with heart failure. Heart failure is defined by the modified Framingham criteria as follow:
  [Major Criteria] 1) Paroxysmal nocturnal dyspnea 2) Orthopnea 3) Neck-vein distension 4) Rales 5) Acute pulmonary edema [Minor Criteria]
  1. Ankle edema
  2. Dyspnea on exertion
  3. Pleural effusion
  4. Tachycardia (HR ≧ 120/min) * For establishing a definite diagnosis of heart failure, 2 Major criteria or 1 major and 2 minor criteria must be present concurrently
Cancer incidence | 5 years
  1. Non-metastatic cancer (not present prior to randomization)
  2. Metastatic cancer (cancer that was metastatic at presentation, metastasis of a non-metastatic cancer presents at baseline, or blood cancer) Non-melanoma skin cancer was excluded cancer end points.
Cancer death | 5 years
  Cancer death is defined as death from cancer cause.
Composite of all-cause mortality, myocardial infarction, ischemic stroke, coronary revascularization, lower extremity revascularization, critical lower extremity ischemia, major bleeding, hospital admission for heart failure, cancer death | 5 years
  Composite of all-cause mortality, myocardial infarction, ischemic stroke, coronary revascularization, lower extremity revascularization, critical lower extremity ischemia, major bleeding, hospital admission for heart failure, cancer death

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, PhD, Principal Investigator — Kyoto University, Graduate School of Medicine
Locations (1):
- Kyoto University Hospital, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: No